CLINICAL TRIAL: NCT00325637
Title: A Multi-Center, Double Blind, Randomized and Non-Inferiority Clinical Study of Cilnidipine to Compare the Effects on Cerebral Blood Flow With Losartan in Patients With Ischemic Stroke Hypertension
Brief Title: Cilnidipine Effect on High Blood Pressure and Cerebral Perfusion in Ischemic Stroke Patients With Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Choi, Jeongeun/Director, Boryung Pharmaceutical Co., Ltd
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNL-BR3-01-02; CHERISH Study
Record Dates: First submitted 2006-05-11; First posted 2006-05-15 (Estimated); Last update posted 2008-12-12 (Estimated); Status verified 2008-12

CONDITIONS: Hypertension; Stroke
Keywords: CHERISH; Ischemic Stroke
MeSH Terms: conditions — Hypertension; Stroke; Ischemic Stroke | interventions — cilnidipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A,1,III (Active Comparator): To compare the effect of cilnidipine (calcium channel blocker) and losartan (angiotension II receptor blocker) on CBF in patients with ischemic stroke
  Interventions: Drug: cilnidipine

INTERVENTIONS:
Drug: cilnidipine — Cilnidipine 10~20mg, qd, po for 4 weeks.
  Other Names: Arms: Losartan, Cilnidipine; Cinalong

SUMMARY:
The purpose of this study is to compare the effect of cilnidipine (a calcium channel blocker) and losartan (an angiotensin II receptor blocker) on cerebral blood flow (CBF) and blood pressure in hypertensive patients with a previous ischemic stroke.

DETAILED DESCRIPTION:
Design: Multi-center, randomized, double-blind, active control, titrated dose, non-inferiority trial

Population Studied: We will prospectively recruit 250 hypertensive patients who had ischemic stroke 2 or more weeks previously and were admitted at 7 centers in the Seoul metropolitan area in South Korea.

Interventions: After a 2-week washout period, all patients will undergo baseline 99mTc-HMPAO single photon emission computed tomography (SPECT), blood pressure evaluation, NIHSS examination, and laboratory test prior to treatment. The patients will be randomized to receive either cilnidipine 10-20mg or losartan 50-100mg once daily for 4 weeks with a target systolic blood pressure of < 140mmHg and diastolic blood pressure of < 90mmHg. After 4-week treatment, all patients will receive follow-up SPECT and blood pressure evaluation. For the quantitative CBF analysis, SPECT will be performed with a single machine in one center.

Outcome Measures: Primary outcome measure is the percentile change of global CBF on SPECT between pre- and post-treatments. Secondary outcome measures include the percentile change of regional CBF, the proportion of patients less than 8.6% decrease of global CBF, and the change of NIHSS score.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke patients with hypertension

Exclusion Criteria:

* Cardioembolic stroke patients
* Severe hypertensive patients
* Secondary hypertensive patients

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2005-01; Primary Completion 2007-07 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
the changes of global cerebral blood flow | from screnning to weeks 4

SECONDARY OUTCOMES:
The percentile change of regional CBF | from screnning to weeks 4
The proportion of patients less than 8.6% decrease of global CBF | from screnning to weeks 4
The change of NIHSS scores | from screnning to weeks 4

CONTACTS AND LOCATIONS:
Overall Officials: Seong H Park, Professor, Principal Investigator — Seoul National University Budang Hospital; Jeong H Rha, Professor, Principal Investigator — Inha University Hospital; Ja S Koo, Professor, Principal Investigator — Eulji General Hospital; Keun S Hong, Professor, Principal Investigator — Inje University Ilsan Paik Hospital; Yong S Lee, Professor, Principal Investigator — Seoul National University Boramae Hospital; Dong W Kang, Assistant Professor, Principal Investigator — Asan Medical Center
Locations (1):
- Seoul National University Budang Hospital, Seongnam-si, Gyeonggi-do, South Korea